CLINICAL TRIAL: NCT04288726
Title: A Phase 1 Study Evaluating the Safety and Activity of Allogeneic CD30 Chimeric Antigen Receptor Epstein-Barr Virus-Specific T Lymphocytes (CD30.CAR-EBVSTs) in Patients With Relapsed or Refractory CD30-Positive Lymphomas
Brief Title: Allogeneic CD30.CAR-EBVSTs in Patients With Relapsed or Refractory CD30-Positive Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-46862 BESTA
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type; Classical Hodgkin Lymphoma
Keywords: CD30-Positive Lymphoma; Hodgkin lymphoma; non-Hodgkin lymphoma; CD30 CAR
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Phase (Experimental): Four dose levels will be evaluated based on safety data from our current study of CD30 CAR T cells. Cohorts of three to six patients will be enrolled at each dose level The dose is based on the number of CD.30 CAR-EBVT-expressing cells administered. The total number of dose levels evaluated will depend upon toxicities experienced. Dose level cohorts will be numbered sequentially.
  * Dose Level 1: 4 × 10^7 CD30.CAR-EBVST cells
  * Dose Level 2: 1 × 10^8 CD30.CAR-EBVST cells
  * Dose Level 3: 4 × 10^8 CD30.CAR-EBVST cells
  * Dose Level 4: 8 × 10^8 CD30.CAR-EBVST cells
  Interventions: Biological: CD30.CAR-EBVST cells

INTERVENTIONS:
Biological: CD30.CAR-EBVST cells — The dose is based on the number of CD30.CAR-expressing cells. In our previous study the highest dose was 2 × 10^8 cells/m2 and we did not reach an MTD. This will be administered as a single infusion of the full dose for each level, which was already shown to be safe in the first 3 patients treated at dose level 3. Since we have not observed any dose limiting toxicities at the current dose level (Dose Level 3 as of June 2022), we propose to include a new higher dose level (8 × 10^8).There will be a gap of 4 weeks between the first and second patient, and between the second and the third patient, on each dose level.
  Other Names: Allogeneic CD30 Chimeric Antigen Receptor Epstein-Barr Virus-Specific T Lymphocytes

SUMMARY:
This study involved patients that have a cancer called diffuse large B cell lymphoma (DLBCL), NK and T cell lymphomas (NK/TL) or classical Hodgkin lymphoma (cHL) (hereafter these 3 diseases will be referred to as lymphoma). Patients lymphoma has come back or not gone away after treatment. Because there is no standard treatment for the patients cancer at this time or because the currently used treatments do not work fully in all cases, the patients are being asked to volunteer in this research study.

In this study the investigators want to test a type of T cell made from a normal donor. The T cells the investigators will use are called Epstein Barr virus (EBV) specific T cells (EBVSTs) and are cells that the investigators have trained in the laboratory to recognize a EBV which is the virus that causes mono or kissing disease. Some patients with lymphoma have EBV in their cancer cells. Researchers have given T cell lines from normal donor EBVSTs to lymphoma patients who have EBV in their lymphoma cells and have seen responses in about half the patients. The cells have have been generated and are frozen in a bank. The cells are called "allogeneic" (meaning the donor is not related to the patient). CD30.CAR in EBV-specific T cells (called allogeneic CD30.CAR-EBVST) from the blood of healthy donors. The investigators are giving the cells to patients with lymphoma cells that express CD30. If the lymphoma cells also express EBV there may be some benefit from targeting both proteins.

The purpose of this study is to find out the highest safe dose of allogeneic CD30.CAR-EBVST cells given following chemotherapy and used to treat lymphoma. The investigators will learn the side effects of CD30.CAR-EBVST cells in patients and see whether this therapy may help lymphoma patients

DETAILED DESCRIPTION:
Earlier, healthy donors gave blood for us to make CD30.CAR-EBVST cells in the laboratory. These cells were grown and frozen and the investigators will select the donor which the investigators think is the best match for the patient. This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose of CD30.CAR-EBVST cells. Once the lower dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 4 dose levels are studied. If the side effects are too severe, the dose will be lowered or the T cell infusion will be stopped. Both the risks and benefits of this study may be dose related. The investigators don't know the best dose that will provide benefit while minimizing the risks.

To enroll on this study, patients will need to have recovered from toxic effects of previous chemotherapy and not be receiving any other investigational agents. Patients cannot have received an investigational cell therapy or vaccine within the past 6 weeks. Patients cannot have received an investigational small molecule drug within the past 2 weeks.

If patients agree to take part in this study, the investigators will ask the patients to adhere to the following study visits and procedure. After patients have signed the consent form, patients are required to come to the hospital for a series of standard medical screening tests, lymphodepletion chemotherapy with cyclophosphamide and fludarabine, infusion with CD30.CAR-EBVST cell treatment and follow-up visits (See details below).

1. Screening tests

   Screening tests include:
   * Blood tests [Human Leukocyte Antigen (HLA) testing] to help us identify the best match for patients from the banked CD30.CAR-EBVST cells.
   * Blood tests for viruses such as human immunodeficiency virus [HIV], human T cell lymphotropic virus [HTLV], hepatitis B virus and hepatitis C virus.
   * Tumor biopsy test to check the status of CD30.

   Once the investigators find that patients are eligible for this study, patients will be called for additional screening tests before treatment day. The screening tests include:
   * Physical examination
   * Vital signs tests to measure temperature, pulse, respiratory rate and blood pressure
   * Blood tests to measure blood cells, kidney and liver functions
   * Urine test
   * Pregnancy test for women of child-bearing potential
   * Measurements of tumor by routine imaging studies
2. Lymphodepletion chemotherapy Several studies suggest that the infused T cells need room to be able to multiply and grow to accomplish their functions and that this may not happen if there are too many other T cells in the blood stream. Because of that, if patients have NOT had a bone marrow or stem cell transplant recently, patients will receive treatment with cyclophosphamide and fludarabine (chemotherapy drugs) before patients receive the CD30.CAR-EBVST cells if patients doctor thinks this is appropriate. This is called "lymphodepletion". These drugs will decrease the numbers of patients own T cells before the investigators inject the CD30.CAR-EBVST cells. Although the investigators do not expect any effect on the patients tumor with the dose that the patients will receive, these drugs are part of many regimens that are used to treat lymphoma.
3. Treatment with CD30.CAR-EBVST cells

   Each patient will receive a total dose of CAR modified T cells according to the following dosing schedule:
   * Dose Level 1: 4 × 10^7 CD30.CAR-EBVST cells
   * Dose Level 2: 1 × 10^8 CD30.CAR-EBVST cells
   * Dose Level 3: 4 × 10^8 CD30.CAR-EBVST cells
   * Dose Level 4: 8 × 10^8 CD30.CAR-EBVST cells

   The CD30.CAR-EBVST cells will be infused via an IV line at the assigned dose. Before patients receive the infusion, they may be given a dose of acetaminophen or anti-histamine (Benadryl for example) to minimize any possible allergic reaction. The infusion of CD30.CAR-EBVST cells will take within 10 minutes. The investigators will follow patients in the clinic after each infusion for up to 3 hours. The patient will need to stay less than 2 hours away from the Medical Center for 4 weeks after the CD30.CAR-EBVST cell infusion so the investigator can monitor them for side effects.
4. Follow-up visits

On follow-up visits after treatment, patients will also receive a series of standard medical tests:

* Physical examination
* Vital sign tests to measure temperature, pulse, respiratory rate and blood pressure
* Blood tests to measure blood cells, kidney and liver functions
* Urine tests (if clinically necessary)
* Pregnancy test for women of child-bearing potential (if clinically necessary)
* Measurements of tumor by routine imaging studies

After infusion of CD30.CAR-EBVST cells,the patients blood will be collected on follow-up visits at week 1, week 2, week 3, week 4, week 6, week 8, every 3 months for 1 year, every 6 months for 4 more years. Blood samples and tumor biopsies will also be periodically collected, based on the patients doctor's discretion for exploratory tests in the laboratory. After 5 years, in the event there is suspected or new cancer is detected, additional blood sample will also be collected for additional tests.

To learn more about the way the CD30.CAR-EBVST cells are working and how long they last in the body, the investigators will draw blood. The total amount of blood collected on any day is about 4-18 teaspoons (18-87 ml). This volume is considered safe but may be decreased if the patients are anemic. Patients blood will be drawn from a central line if participants have one. The total blood drawn during the patients participation in this study will not exceed 110 teaspoons (546 ml).

The investigators will also look at any scans or biopsies patients have had as standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis and clinical course falling into one of the following categories:

   1. Hodgkin lymphoma
   2. Aggressive non-Hodgkin lymphoma
   3. ALK-negative anaplastic T cell lymphoma or other peripheral T-cell lymphoma
   4. ALK-positive anaplastic T cell lymphoma
2. CD30-positive tumor as assayed in a CLIA certified Pathology Laboratory.
3. Age 12 to 75.
4. Bilirubin 2 times (or 3 times if the patient has Gilbert syndrome) or less than the upper limit of normal.
5. AST 3 times or less than the upper limit of normal.
6. Estimated GFR > 70 mL/min.
7. Pulse oximetry of > 90% on room air
8. EKG shows no significant arrhythmias
9. Karnofsky or Lansky score of > 60%.
10. Available allogeneic T cells with ≥15% expression of CD30CAR determined by flow-cytometry.
11. Recovered from all acute non-hematologic toxic effects of all prior chemotherapy.
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
13. Informed consent explained to, understood by and signed by patient or guardian. Patient or guardian given a copy of the informed consent form.

Exclusion Criteria:

1. Received an investigational cell therapy or vaccine within the past 6 weeks.
2. Received an investigational small molecule drug within the past 2 weeks.
3. Received CD30 antibody-based therapy within the previous 4 weeks.
4. Received gemcitabine-containing chemotherapy within the previous 12 weeks
5. History of hypersensitivity reactions to murine protein-containing products.
6. Pregnant or lactating.
7. Tumor in a location where enlargement could cause airway obstruction (determined at the investigators' discretion).
8. Current use of systemic corticosteroids at a dose equivalent to higher than 10 mg/day of prednisone.
9. Active significant, uncontrolled bacterial, viral or fungal infection.
10. Symptomatic cardiac disease (NYHA Class III or IV disease).

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2037-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rate (DLT) by CTCAE 5.0 | 28 days
  Any Grade 5 event, / Non-hematologic dose-limiting toxicity is any Grade 3 or Grade 4 non-hematologic toxicity that affects the cardiopulmonary system, or corresponds to neurotoxicity, or otherwise fails to return to Grade 2 within 72 hours, / Grade 2-4 allergic reaction to T-Cells, / Grade 3-4 GVHD, / Hematologic dose limiting toxicity is defined as any Grade 4 hematologic toxicity that fails to return to Grade 2 or baseline (whichever is more severe) within 14 days or within 28 days for patients with evidence of bone marrow disease.

SECONDARY OUTCOMES:
Rate of Anti-Tumor effect Objective Response (OR) | 6 to 8 weeks post CTL infusion
  Objective response rate is defined as complete response and partial response
Duration of response | Up to 5 years
  Response duration will be measured from the time of initial response until documented tumor progression.
Stable disease (SD) rate | 6 to 8 weeks post CTL infusion
  SD will be defined as the proportion of patients that have stable disease
Duration of SD | Up to 5 years
  Stable disease is measured from the start of the treatment until the criteria for progression are met.
Progression free survival (PFS) | Up to 5 years
  PFS is defined as the time from treatment until objective tumor progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No